CLINICAL TRIAL: NCT06644586
Title: COMPARISON of VIDEO LARYNGOSCOPY and MACINTOSH LARYNGOSCOPY in PEDIATRIC PATIENTS UNDERGOING ELECTIVE SURGERY
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Elzem SEN, Gaziantep University, University of Gaziantep
Other Study IDs: 2022/100
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Patients Undergoing Operation
Keywords: video laryngoscopy; direct laryngoscopy; pediatric patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: videolaryngoscopy — The patients intubated with video laryngoscopy
Other: Direct Laryngoscopy — The patients intubated with direct laryngoscopy

SUMMARY:
In this study, we aimed to observe the intubation conditions in patients using Endolarenx video laryngoscope and Macintosh Blade in laryngoscopy to identify the advantages and disadvantages of using video laryngoscopy in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* One hundred pediatric patients, aged under 18 years, weighing between 10-40 kg, and classified as American Society of Anesthesiologists (ASA) I-II-III risk group

Exclusion Criteria:

* Patients with congenital airway deformities, patients with known or predicted difficult intubation, patients undergoing emergency surgery, patients classified above ASA III, and patients whose parents did not consent were excluded from the study

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who underwent elective surgery at Gaziantep University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mean intubation time | The time from the entry of the laryngoscope into the oral cavity until the appearance of the EtCO2 trace on the capnograph.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided